CLINICAL TRIAL: NCT06156501
Title: Psychological Factors Influencing the Patient-reported and Functional Outcome of ACL Reconstruction and Their Sex-specific Differences
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lorenz Pichler, MD, Resident Doctor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100391
Record Dates: First submitted 2023-11-15; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: ACL Tear
Keywords: Psychology; Gender Medicine
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACL Reconstruction (Experimental): Patients undergoing ACL reconstruction
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: ACL Reconstruction — Reconstruction of the anterior cruciate ligament

SUMMARY:
Psychological parameters among patients undergoing ACL reconstruction and their impact on the patient-reported and functional outcome of reconstruction will be prospectively evaluated

ELIGIBILITY:
Inclusion Criteria:

* ACL tear
* Over 18 years
* Patient information and consent
* No preexisting knee conditions prior ACL tear;

Exclusion Criteria:

* Under 18 years
* Preexisting knee conditions
* Accompanying knee injuries apart from ACL tear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Knee Function (Lysholm Knee Score, Points) | 0 to 12 months after surgery
  Established patient-reported knee related score
Objective Knee Function | 0 to 12 months after surgery
  Standardized physiotherapeutical return to sports test battery, (pass/no pass)
Psychological Status (ACL-RSI, points) | 0 to 12 months after surgery
  Established psychological self-awareness score
Patient Pain (Visual Analoge Scale (points) | 0 to 12 months after surgery
  Patient reported pain

SECONDARY OUTCOMES:
Graft Maturation | 6 months postoperative
  Knee MRI assessing graft maturation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria